CLINICAL TRIAL: NCT05124314
Title: Comparison of Efficacy and Safety of Sequential Use of Mifepristone and Misoprostol vs Misoprostol Alone in Women With Early Pregnancy Loss: Randomized Controlled Trial
Brief Title: Comparison of Two Different Drug Regimens for Medical Treatment of Early Pregnancy Loss
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Hospital Merkur (Other)
Collaborators: University of Zagreb School of Medicine (Unknown)
Responsible Party: Principal Investigator, Mate Milas, Principal Investigator, Clinical Hospital Merkur
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0001
Record Dates: First submitted 2021-10-25; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Abortion, Missed
Keywords: Missed miscarriage; Mifepristone; Misoprostol; Medical management
MeSH Terms: conditions — Abortion, Missed; Abortion, Incomplete | interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Intervention Model Description: A randomized, parallel group, single center study. Before receiving vaginal misoprostol (800 mcg, repeated after 24 hours if no pregnancy tissue is lost), patients will be randomized to either oral mifepristone (600 mg) or nothing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mifepristone and Misoprostol (Experimental): Patients receive oral mifepristone (600 mg) 48 hours before medical treatment with vaginal misoprostol (800 mcg repeated after 24 hours if no pregnancy tissue is lost).
  Interventions: Drug: Mifepristone, Oral, 200 Mg; Drug: Misoprostol Pill
- Misoprostol (Active Comparator): Medical treatment with vaginal misoprostol (800 mcg repeated after 24 hours if no pregnancy tissue is lost).
  Interventions: Drug: Misoprostol Pill

INTERVENTIONS:
Drug: Mifepristone, Oral, 200 Mg — Adding 600 mg of oral Mifepristone to the regular treatment with vaginal Misoprostol 800 mcg
  Other Names: Mifegyne
  Arms: Mifepristone and Misoprostol
Drug: Misoprostol Pill — Regular treatment with vaginal Misoprostol 800 mcg
  Other Names: Mispregnol

SUMMARY:
The purpose of this study is to compare the safety and efficacy of a combination of two drugs (mifepristone and misoprostol) to only one of these drugs (misoprostol) in medical management of missed miscarriage up to 13+6 weeks of pregnancy (early pregnancy loss).

The investigators aim to enroll 220 patients within two years which would be enough to determine the difference between these two treatments with confidence.

DETAILED DESCRIPTION:
Aim: To investigate the safety and efficacy of combination of mifepristone and misoprostol versus misoprostol alone in medical management of early pregnancy loss.

Primary objective: To test the hypothesis that the sequential combination of mifepristone and misoprostol is superior to misoprostol alone for the complete evacuation of uterus in patients diagnosed with early pregnancy loss.

Secondary objectives: To test the hypothesis that the addition of mifepristone reduces the need for further doses of misoprostol, duration of bleeding, complication rate and side effect frequency. The investigators will also evaluate if the addition of mifepristone improves patient satisfaction and quality of life.

Women with a diagnosis of early pregnancy loss that opt for medical treatment and sign an informed consent will be included. The participants will be randomized to two groups. First group will receive oral mifepristone (600 mg) and the second group will not. The remaining course of treatment will be the same for both groups including giving misoprostol (800 mcg vaginally) 48 hours after receiving mifepristone for the first group or immediately for the second group. 24 hours after receiving first dose of misoprostol, one more dose of misoprostol (also 800 mcg vaginally) will be given if no pregnancy tissue is lost.

Three weeks after medical treatment, primary and secondary outcomes will be assessed. In case of unsuccessful treatment (incomplete evacuation of uterus), surgical evacuation will be performed.

220 women will be randomized in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with missed miscarriage in the first 13+6 weeks of pregnancy opting for medical management
* Age 18 years and older
* Intra-uterine pregnancy
* Hemodynamically stable patient
* No signs of infection
* No signs of incomplete miscarriage
* Willing and able to give informed consent

Exclusion Criteria:

* Women opting for alternative methods of miscarriage management (expectant or surgical)
* Diagnosis of incomplete miscarriage
* Life threatening bleeding
* Hemodynamically unstable patient
* Contraindications to mifepristone or misoprostol use for example chronic adrenal failure, known hypersensitivity to either drug, haemorrhagic disorders and anticoagulant therapy, prosthetic heart valve or history of endocarditis, existing cardiovascular disease, severe asthma uncontrolled by therapy or inherited porphyria
* Previous participation in this trial
* Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete evacuation of uterus | Three weeks after randomization
  Complete evacuation of uterus will be assessed by clinical and ultrasound examination three weeks after treatment. There should be no vaginal bleeding and no suspicion of retained products of conception on ultrasound scan (endometrial thickness <= 15 mm) to declare the treatment successful.

SECONDARY OUTCOMES:
Total misoprostol dose used | Up to three weeks after randomization
  Total dose of misoprostol used during treatment
Complications | Up to three weeks after randomization
  Frequency of complications (by type)
Side effects | Up to three weeks after randomization
  Type and degree of side effects experienced as reported in the patient's diary
Duration of vaginal bleeding | Up to three weeks after randomization
  Duration of vaginal bleeding as reported in the patient's diary
Hemoglobin change | At randomization and three weeks after randomization
  Hemoglobin change from randomization until three weeks after treatment
Patient quality of life | At randomization, 24 hours after taking first misoprostol dose and three weeks after randomization
  Overall health status measured using EuroQol-5 dimensions-5 levels questionnaire's (EQ-5D-5L) VAS (visual analog scale) score ranging from 0 to 100 where 0 represents worst health the participant can imagine and 100 represents the best health the participant can imagine
Patient satisfaction | Three weeks after randomization
  Overall patient satisfaction with the treatment measured using validated paper-based Client Satisfaction Questionnaire (CSQ-8) score ranging from 4 to 32, where higher number represents higher satisfaction
Indication for surgical treatment | Three weeks after randomization
  Type and incidence of indications for surgical evacuation of uterus in case of unsuccessful medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mate Milas, MD, Principal Investigator — Clinical Hospital Merkur
Locations (1):
- Clinical Hospital Merkur, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No